CLINICAL TRIAL: NCT01797562
Title: Clinical Evaluation of T.R.U.E. Test Panel 3.2 in Children and Adolescents (PREA II)
Brief Title: Clinical Evaluation of T.R.U.E. Test Allergens in Children an Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP 12 7NEW 401
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-04

CONDITIONS: Allergic Contact Dermatitis
Keywords: Contact dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Allergic Contact; Dermatitis, Contact; Eczema

STUDY DESIGN:
Intervention Model Description: 3 T.R.U.E. Test panels were applied to the paraspinal regional of the back and were to be worn for approximately 48 hours. Post application evaluations were performed at days 3, 4, 7(+1) and 21(+2).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Response Rates: 7 new and 4 reformulated allergens (Experimental): Subjects will be patched with TRUE Test Panels 1.3, 2,2 and 3.2. Panel 1 allergens nickel sulfate (0.60 mg/cm2), potassium dichromate (0.054 mg/cm2), fragrance mix (0.050 mg/cm2) and ethylenediamine dihydrochloride (0.050 mg/cm2), Panel 2 allergen Methyldibromoglutaronitrile (0.0053 mg/cm2) and Panel 3 allergens Gold sodium thiosulfate (0.075 mg/cm2), Hydrocortisone-17-butyrate (0.020 mg/cm2), Bacitracin (0.60 mg/cm2), Parthenolide (0.0030 mg/cm2), Disperse blue 106 (0.050 mg/cm2 in PVP), 2-Bromo-2-nitropropane-1,3-diol (Bronopol) (0.25 mg/cm2) will be evaluated
  Interventions: Diagnostic Test: Panels 1.3, 2.2 and 3.2 experimental allergens

INTERVENTIONS:
Diagnostic Test: Panels 1.3, 2.2 and 3.2 experimental allergens — Three allergen panels will be applied to the upper backs of study subjects and will be worn for 48 hours. Allergen test sites will be evaluated at 3, 4, 7(±1) and 21(±2) days post application.

SUMMARY:
The objective of the study was to evaluate the diagnostic performance and safety of T.R.U.E. Test allergens in pediatric subjects aged 6-17 years old. In total, 11 allergens were evaluated; 7 new allergens on panels 2.2 and 3.2 and 4 previously approved allergens for which changes were made to dose and excipient.

DETAILED DESCRIPTION:
The evaluation of 7 new allergens on panels 2.2 and 3.2, Gold sodium thiosulfate, Hydrocortisone-17-butyrate, Bacitracin, Parthenolide, Methyldibromoglutaronitrile, Disperse blue 106, and Bronopol was the original objective of the study. The protocol was amended to include evaluation of 4 reformulated allergens; neomycin sulfate, potassium dichromate, ethylenediamne dihydrochloride and fragrance mix.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and history potentially consistent with allergic contact dermatitis
* Children and adolescents 6-17 years of age, in general good health
* Adolescent females 15 years of age or older (or with menarche) must consent to a urine pregnancy test; urine test results must be negative for study inclusion
* Informed consent must be signed and understood by subject. If underage, informed consent must be signed and understood by parent or legal guardian, consistent with all institutional, local and national regulations

Exclusion Criteria:

* Topical corticosteroid treatment during the last 7 days on or near the test area.
* Systemic treatment with corticosteroids or other immunosuppressives during the last 7 days.
* Subjects currently receiving (or received during the previous 3 weeks) other investigational drugs, treatments or devices, or participating in another clinical study
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks
* Acute dermatitis outbreak or dermatitis on or near the test area on the back
* Subjects unable to comply with activity restrictions (e.g. protecting test panels from excess moisture due to showering or vigorous activity)
* Subjects unable or unwilling to comply with multiple return visits
* Female subjects 15 years of age (or with onset of menarche) and older unable to consent to a urine pregnancy test, or those with a positive pregnancy test

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2015-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory Dunnick, MD, Principal Investigator — Anschutz Health and Wellness Center, University of Colorado, Aurora, CO; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, Louisville, KY; Lawrence Eichenfield, MD, Principal Investigator — Rady Children's Hospital, San Diego; Patricia Norris, MD, Principal Investigator — Oregon Health and Science University
Locations (4):
- United States (4):
  - Rady Children's Hospital, San Diego, California
  - Anschutz Health and Wellness Center, University of Colorado, Aurora, Colorado
  - Dermatology Specialists, Louisville, Kentucky
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from patients visiting dermatology, allergy or similar medical practices and clinics, and who are likely to require diagnostic patch testing. Study subjects must be otherwise healthy, and fulfill entry criteria.
Pre-assignment Details: Entry criteria required avoidance of systemic or topical (near the test area) corticosteroid treatment during the 7 days prior to patch application, and any treatment with UV light for 3 weeks prior to patch application.
Groups:
- Evaluation of T.R.U.E. Test Experimental Allergens: 11 experimental patch test allergens:0.60mg/cm2 neomycin, 0.054 mg/cm2 potassium dichromate, 0.50 mg/cm2 fragrance mix, 0.050 mg/cm2 ethylenediamine, 0.075 mg/cm2 gold,0.020 mg/cm2 hydroxycortisone, 0.60 mg/cm2 bacitracin, 0.0030 mg/cm2 parthenolide,0.050 mg/cm2 disperse blue and 0.25 mg/cm2 bronopol were applied to the skin for 48 hours.
Period: Overall Study
Arm/Group | Evaluation of T.R.U.E. Test Experimental Allergens
Started | 116
Completed | 111
Not Completed | 5
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Arm/Group | Positive Response Rates: 7 New and 4 Reformulated Allergens
Number analyzed (Participants) | 116
Age, Continuous [Mean (Full Range); unit: years] | 12.6 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 78
  More than one race | 12
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative, Positive, Irritant or Doubtful Reaction Scores
Description: Reactions at patch test sites were evaluated:Negative: No reaction, Irritant: Discrete, patchy, follicular, or homogenous erythema with no infiltration, Doubtful: Faint macular or homogenous erythema with no infiltration, 1+: Faint macular or homogenous erythema with no infiltration, 2+: Erythema, papules, infiltration, discrete vesicles 3+: Coalescing vesicles, bullous reaction
Time Frame: Investigator Determination of Positive Reaction: 21 days post application
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Response Rates: 7 New and 4 Reformulated Allergens
Number analyzed (Participants) | 111
Participants
  Neomycin sulfate: Negative | 49
  Neomycin sulfate: Positive | 3
  Neomycin sulfate: Irritant | 0
  Neomycin sulfate: Doubtful | 1
  Neomycin sulfate: Not Tested with this Allergen | 58
  Potassium dichromate: Negative | 50
  Potassium dichromate: Positive | 2
  Potassium dichromate: Irritant | 0
  Potassium dichromate: Doubtful | 1
  Potassium dichromate: Not Tested with this Allergen | 58
  Fragrance Mix: Negative | 48
  Fragrance Mix: Positive | 2
  Fragrance Mix: Irritant | 0
  Fragrance Mix: Doubtful | 3
  Fragrance Mix: Not Tested with this Allergen | 58
  Ethylenediamine: Negative | 53
  Ethylenediamine: Positive | 0
  Ethylenediamine: Irritant | 0
  Ethylenediamine: Doubtful | 0
  Ethylenediamine: Not Tested with this Allergen | 58
  MDBGN: Negative | 107
  MDBGN: Positive | 1
  MDBGN: Irritant | 0
  MDBGN: Doubtful | 3
  MDBGN: Not Tested with this Allergen | 0
  Gold: Negative | 69
  Gold: Positive | 31
  Gold: Irritant | 0
  Gold: Doubtful | 11
  Gold: Not Tested with this Allergen | 0
  Hydrocortisone: Negative | 106
  Hydrocortisone: Positive | 2
  Hydrocortisone: Irritant | 0
  Hydrocortisone: Doubtful | 3
  Hydrocortisone: Not Tested with this Allergen | 0
  Bacitracin: Negative | 90
  Bacitracin: Positive | 16
  Bacitracin: Irritant | 0
  Bacitracin: Doubtful | 5
  Bacitracin: Not Tested with this Allergen | 0
  Parthenolide: Negative | 97
  Parthenolide: Positive | 7
  Parthenolide: Irritant | 0
  Parthenolide: Doubtful | 7
  Parthenolide: Not Tested with this Allergen | 0
  Disperse Blue: Negative | 102
  Disperse Blue: Positive | 4
  Disperse Blue: Irritant | 0
  Disperse Blue: Doubtful | 5
  Disperse Blue: Not Tested with this Allergen | 0
  Bronopol: Negative | 89
  Bronopol: Positive | 19
  Bronopol: Irritant | 0
  Bronopol: Doubtful | 3
  Bronopol: Not Tested with this Allergen | 0

2. Secondary Outcome: Number of Participants With Late or Persistent Positive Patch Test Reactions
Description: Late reactions are positive reactions that initially occur at 7-21 days after application of the panels.
  Persistent reactions are positive reactions that persist from one visit to the next.
  Numbers reported only include late or persistent positive patch test reactions. Not all positive reactions are late or persistent.
Time Frame: Day 7-21
Population: Per protocol population consisted of all subjects who were applied with all panels, whose panels remained in place for approximately 48 hours and returned for all visits.
Measure: Count of Participants; unit: Participants
Groups:
- Evaluation of T.R.U.E. Test Experimental Allergens: Percentage of positive patch test results will be reported for 11 experimental allergens tested in a pediatric population
Arm/Group | Evaluation of T.R.U.E. Test Experimental Allergens
Number analyzed (Participants) | 111
Participants
  Neomycin sulfate: Persistent Reactions | 2
  Neomycin sulfate: Late Reactions | 1
  Neomycin sulfate: Neither | 108
  Potassium dichromate: Persistent Reactions | 0
  Potassium dichromate: Late Reactions | 1
  Potassium dichromate: Neither | 110
  Fragrance mix: Persistent Reactions | 2
  Fragrance mix: Late Reactions | 0
  Fragrance mix: Neither | 109
  Ethylenediamine: Persistent Reactions | 0
  Ethylenediamine: Late Reactions | 0
  Ethylenediamine: Neither | 111
  MDBGN: Persistent Reactions | 0
  MDBGN: Late Reactions | 1
  MDBGN: Neither | 110
  Gold: Persistent Reactions | 15
  Gold: Late Reactions | 15
  Gold: Neither | 81
  Hydrocortisone: Persistent Reactions | 0
  Hydrocortisone: Late Reactions | 2
  Hydrocortisone: Neither | 109
  Bacitracin: Persistent Reactions | 9
  Bacitracin: Late Reactions | 7
  Bacitracin: Neither | 95
  Parthenolide: Persistent Reactions | 1
  Parthenolide: Late Reactions | 6
  Parthenolide: Neither | 104
  Disperse Blue: Persistent Reactions | 2
  Disperse Blue: Late Reactions | 2
  Disperse Blue: Neither | 107
  Bronopol: Persistent Reactions | 6
  Bronopol: Late Reactions | 13
  Bronopol: Neither | 92

ADVERSE EVENTS:
Time Frame: Days 2-21
Description: Adverse events cannot be attributed to a single allergen as the allergen panels contained all allergens.
Groups:
- Evaluation of T.R.U.E. Test Experimental Allergens: Adverse events were captured for subjects patched with TRUE Test Panels 1.3, 2,2 and 3.2. Panel 1 allergens nickel sulfate (0.60 mg/cm2), potassium dichromate (0.054 mg/cm2), fragrance mix (0.050 mg/cm2) and ethylenediamine dihydrochloride (0.050 mg/cm2), Panel 2 allergen Methyldibromoglutaronitrile (0.0053 mg/cm2) and Panel 3 allergens Gold sodium thiosulfate (0.075 mg/cm2), Hydrocortisone-17-butyrate (0.020 mg/cm2), Bacitracin (0.60 mg/cm2), Parthenolide (0.0030 mg/cm2), Disperse blue 106 (0.050 mg/cm2 in PVP), 2-Bromo-2-nitropropane-1,3-diol (Bronopol) (0.25 mg/cm2) will be evaluated
Arm/Group | Evaluation of T.R.U.E. Test Experimental Allergens
Serious Adverse Events (participants affected / at risk) | 1/116
Other Adverse Events (participants affected / at risk) | 47/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evaluation of T.R.U.E. Test Experimental Allergens (N=116)
Appendicitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evaluation of T.R.U.E. Test Experimental Allergens (N=116)
Chest pain (General disorders) | 1 (1) — Chest pain
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Discomfort (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6)
Pain (General disorders) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9)
Pyoderma (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No